CLINICAL TRIAL: NCT02984007
Title: Addressing Vaccine Hesitancy: Pan-Canadian Validation of an Effective Strategy
Brief Title: PROMOtion of VAccination in Canada (PromovaC Study)
Acronym: PromovaC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: University of British Columbia (Other); University of Toronto (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Arnaud Gagneur, Principal Investigator, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-1578
Record Dates: First submitted 2016-11-30; First posted 2016-12-06 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Vaccination Promotion
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Educational session based on the motivational interviewing
  Interventions: Behavioral: Motivational Interviewing
- Information flyer (Other): Information flyer on childhood vaccines
  Interventions: Other: Information flyer

INTERVENTIONS:
Behavioral: Motivational Interviewing — Mothers randomized in the intervention group will receive an educational session based on the motivational interviewing (MI) approach with a research assistant (RA). The RA will have first received a standardized training session on the content and techniques of MI.
  The MI intervention will be carried out in simple and understandable language in order to allow discussion and questions from parents rather than provide prescriptive and direct information. The intervention will last approximatively 15 to 20 minutes.
  Arms: Motivational Interviewing
Other: Information flyer — Mothers randomized in the control group will receive a locally information flyer on childhood vaccines without any oral explanation by the research assistant.
  Arms: Information flyer

SUMMARY:
Synopsis: In most countries, there is an increase in the number of parents who refuse some, most or all vaccines or who adopt delayed vaccination schedule. Vaccine hesitancy (VH) is a global phenomenon that needs to be measured and addressed. However, to this date, no effective strategy has been identified. Dr Gagneur have developed and validated a new approach to educate parents of newborns about vaccination, based on motivational interviewing (MI) techniques. MI is a method to elicit and strengthen motivation for change based on the person's own arguments for change that has been shown effective for the adoption of many preventive health behaviors. This approach has been validated for vaccination during a pilot study as well as in a provincial RCT in Quebec. Now that a proof of concept has been made in Quebec, the investigators will validate the approach in other contexts (e.g. English-speaking provinces and settings with different ways to deliver maternity care and childhood vaccines).

Hypothesis: An educational strategy, based on MI techniques, delivered in the maternity ward increases parents' intention to vaccinate their infant, reduces VH scores and increases infants' vaccine uptake in Quebec. This approach may be applicable across the country in order to tackle VH and thus improve infants' vaccine coverage (VC).

Objective: To evaluate the impact of the MI intervention on parents' intention to vaccinate their child and their VH score and on infants' VC at 3 months of age, in a pan-Canadian context.

Methods: Multicentre RCT in maternity wards of 5 provinces (QC, BC, ON, NS/PE). Parents will be randomized to receive the MI intervention (intervention group) or to receive an information flyer on vaccines (control group). MI intervention will be delivered by research assistant that will have first received a standardized training session on the content and techniques of MI. Parents will complete a self-administered questionnaire to measure knowledge and vaccination intention as well as VH before and after the intervention. Immunization data will be collected through an online questionnaire sent when the child will reach 3 months of age.

Expected benefits: The strategy will be validated across different immunization programs from 5 Canadian provinces to take account of the differences in logistics and cultural contexts. Results from this study will provide to the provincial and national public health authorities an effective strategy to tackle VH.

DETAILED DESCRIPTION:
OBJECTIVES

Main objective: To evaluate the impact of the motivational interviewing (MI) intervention on parents' intention to vaccinate their infant and their vaccine hesitancy (VH) score in a Pan-Canadian context. In order to explore differences in the intervention's impact according to cultural and organizational factors, all analysis will also be conducted at the level of each center.

Specific objectives:

1. To assess parents' intention to vaccinate their infant before the intervention and immediately after the intervention, globally and at each center level.
2. To assess parents' VH scores before the intervention, immediately after the intervention and when their infant is 3 months of age, globally and at each center level.
3. To assess parents' knowledge, attitudes and beliefs (KAB) about vaccination before the intervention, immediately after the intervention and when their infant is 3 months of age:

   * Descriptive analysis according to a composite model inspired from the Health Belief Model (HBM), the Theory of Planned Behavior, and the VH measures (based on a validated questionnaire);
   * Research of the determinants of vaccination intention.
4. To compare vaccine coverage (VC) at 3 months of age of infants whose parents has received (intervention group) or not (control group) the intervention in the maternity ward during the recruitment period.

STUDY DESIGN

This study is a multicentre randomized controlled trial (RCT) with single unit of randomization that will be conducted in maternity wards of 5 provinces: Quebec (QC), British Columbia (BC), Ontario (ON), and Nova Scotia (NS)/ Prince Edward Island (PEI). In each center, parents will be randomized to receive the MI intervention (intervention group) or to receive an information flyer on childhood vaccines (control group). The flyer that will be given to mothers of the control group will be the one that is usually given to parents at the maternity ward or at the first home visit after birth during the first week. Thus, flyers will be different according to the participating regions in this study. Randomization will be stratified by center and will be made in blocks of 4, 6 and 8 participants.

STUDY POPULATION

Study participants

The study population will include 1,600 mothers of infants born in the participating maternity wards during the recruitment period.

Study centers

The study will be conducted in 6 maternity wards located in 4 different centers:

1. Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, QC;
2. B.C. Women's Hospital & Health Centre, Vancouver, BC and Surrey Memorial Hospital, Surrey, BC;
3. North York General Hospital, Toronto, ON;
4. IWK Health Centre, Halifax, NS and Queen Elizabeth Hospital, Charlottetown, PE.

The choice of these 6 maternity wards is the best compromise between the study feasibility and the diversity of the Canadian population. More than 2,500 deliveries per year occur in each maternity ward (except for Queen Elizabeth Hospital with approximately 1200 annual births), which ensures the feasibility of the study.

CONDUCT OF STUDY

Enrollment

Each subject must participate in the informed consent process and sign and date the informed consent form before any procedures specified in this protocol are performed. Mothers attending the participant maternity wards will be entirely free to participate in the study. Benefits of the study will be the chance for the parents to discuss childhood immunizations in a non-confronting and non-judgemental climate and the improvement of their knowledge. Participation in the study will not involve risk, besides the risk of breach of confidentiality for which precautions will be taken.

Regulatory considerations

The study will be registered with ClinicalTrials.gov.

Recruitment

Mothers will be approached to participate during the postpartum stay at the maternity ward. The MI intervention will be delivered by a research assistant (RA) (or a research nurse) that will have first received a standardized training session on the content and techniques of MI. Since the postpartum stay may last less than 24 hours in some provinces, RAs will recruit mothers in a chronological way according to the birth time of the mother to ensure to meet the highest number of mothers as possible.

The recruitment will be conducted during 4 to 6 months. In the Quebec RCT, 25 participants were recruited in average each week, so it is feasible to recruit 400 participants within 4 to 6 months.

Study plan

After the mothers agree to participate, they will have to complete an initial questionnaire (Q1) to assess their intention to vaccinate, their VH scores and their KAB about vaccination, as well as their socio-demographics characteristics. RAs will collect this questionnaire and proceed to the randomization of the participating mother to receive the MI intervention or to receive a flyer on childhood immunizations. Depending on the randomization result, RAs will perform the MI intervention with the parents or only give the information flyer. RAs will then distribute a similar questionnaire (Q2) to parents of both groups to assess their intention to vaccinate, their VH scores and their KAB about vaccination, as well as their satisfaction of the intervention received (MI or flyer). Before leaving the maternity ward, parents will have to return their completed questionnaire to the RA or in a designated place. When the child is 3 months of age, an online survey (Q3) will be sent to participants by email to assess their VH score and their KAB as well as the child's vaccine status.

Standardization of the intervention

To ensure that the content of the information sessions will be standardized and similar for each center or RA, a reference document on the primary vaccination (vaccines administered before the age of 1 year) will be made according to the provincial recommendations for each center and will be used for the training of RAs. This training will be conducted over 3 days including supervision via audio recordings (2 days + 1 day). First, RAs will participate in a 2-day centralized training seminar in Montreal on the MI techniques given by a certified trainer before the beginning of the study. Subsequently, RAs will practice their MI skills during a 4 to 6-week trial period in their respective maternity ward. During this time, RAs will send an online audio recording of their MI intervention with a mother in the maternity ward (a separate informed consent form will be signed by these mothers to authorize the record and the sending of the MI intervention). The audio recordings will be securely transferred to the certified MI trainer through a web-based application named REDCap (Research Electronic Data Capture). Based on this recording, the certified MI trainer will assess their MI skills and offer them support and feedback to improve their practice. After 6 weeks of trial, the study coordinator and the certified MI trainer will visit each center to give individual feedback and coaching to each RA. They will observe and validate the MI intervention performed by the RAs and identify possible barriers to the implementation of the study according to each maternity ward. This training framework is consistent with the literature since MI training indeed requires training in 2 steps with feedback training and coaching in real situations after the initial training. Data collected during the 6-week trial period will be discarded since the RAs will be practising conducting the study. Data will only be used to monitor good clinical practices (GCPs) in each center during the audit by the study coordinator. After this training, RAs will officially start the recruitment in the maternity wards. The MI trainer will be available to answer questions and offer support to the RAs regarding their MI techniques throughout the study.

Confidentiality protection

Source documents containing names, addresses and other contact information of participants will be stored at each local site in individual folders, identified by the assigned participant identification number (PID) number. These documents are stored in locked filing cabinets in a secure research facility, with controlled access, limited to authorized staff and investigators. No personal identifiers will appear in any summary or report of the study data and will not be sent to the coordinating center.

STATISTICAL CONSIDERATIONS

Sample size

In order to identify a statistically significant amelioration of 8% in parents' intention to vaccinate, and taking account of a basic intention to vaccinate of 78%, a risk of alpha error of 0.05 and a power of 80%, a total of 400 parents by center will be included. This sample size will also allow detect a minimum of 5% reduction in VH scores in each center. The total sample of 1,600 families will allow detecting a significant amelioration of 6% in infants' VC.

Data analysis

A descriptive analysis of responses from Q1, Q2 and Q3 will be conducted. Q1 and Q2 responses as well as Q1 and Q3 responses (KAB, vaccination intention and VH scores) will be compared for mothers belonging to the intervention group in order to assess intervention's effectiveness, globally and for each participating center. Q1, Q2 and Q3 responses (KAB, vaccination intention and VH scores) will be also compared between intervention and control groups in order to demonstrate the MI intervention's effectiveness compared to the information flyer. Parents' intention to vaccinate their infant measured before the intervention will be dichotomized as "certainly" vs. "probably"; "probably not" and "certainly not" and compared to all covariates measured before the intervention. Multivariate logistic regression analysis will be conducted to identify independent determinants influencing vaccination intention. Regarding VC, it will be defined as the proportion of children having a complete vaccine status on the total of participating children. A child is considered having a complete vaccine status if he has received all vaccines and antigens recommended by his respective provincial immunization schedule at 3 months of age.

Q1 and Q2 responses (KAB, vaccination intention and VH scores) will be first compared using McNemar's test and Wilcoxon's signed rank test for paired data for mothers belonging to the intervention group. Thereafter, Q1, Q2 and Q3 responses (KAB, vaccination intention and VH scores) will be compared between intervention and control groups using the Chi-square test or the Fisher's exact test as appropriate while continuous variables will be compared using the Student's t-test or the Mann-Whitney U test as appropriate. Moreover, covariates will be compared with vaccination intention using the appropriate tests mentioned. In multivariate analysis, collinearity of the variables included in the model will be checked and the model adequacy will be assessed by the Hosmer-Lemeshow test and the deviance test. Finally, VC will be analyzed globally, comparing proportion of properly vaccinated children between intervention and control groups using the Chi-square test. The SAS software (version 9.4, SAS Institute, Inc., Cary, NC) will be used for all statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* All mothers of infants born in 1 of the 6 participating maternity wards.

Exclusion Criteria:

* Mothers aged <18 years;
* Mothers who do not speak English or French;
* Any health situation of the newborn or the mother requiring acute care (i.e. if the newborn needs to be hospitalized in the neonatology unit or if the mother has an incompatible condition for an interview);
* Mothers who have participated in one of the two studies evaluating the impact of the MI intervention in the Eastern Townships in 2009-2010 and in the province of Quebec in 2014-2015.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Vaccination status of the child at 3 months of age | 3 months after the intervention at the maternity ward
  Information on the first vaccines that the child might have received assessed at 3 months of age by an online questionnaire sent to parents by email.

SECONDARY OUTCOMES:
Intention to vaccinate | During the 24-hour postpartum stay at the maternity ward
  Parents' intention to vaccinate their child at 2 months of age assessed by a questionnaire based on the Health Belief Model (HBM) before and after the intervention at the maternity ward.
Vaccine hesitancy | During the 24-hour postpartum stay at the maternity ward and 3 months later at home
  Parents' vaccine hesitancy score assessed by a questionnaire based on the Parent Attitudes about Childhood Vaccines (PACV) before and after the intervention at the maternity ward and 3 months later at home.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Gagneur, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (6):
- Canada (6):
  - Surrey Memorial Hospital, Surrey, British Columbia
  - B.C. Women's Hospital & Health Centre, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - North York General Hospital, Toronto, Ontario
  - Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Centre hospitalier universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No